CLINICAL TRIAL: NCT00268697
Title: A Double-Blind, Double-Dummy, Randomized, Parallel Group, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 100 mg and Lapaquistat Acetate 100 mg Administered in Combination With Ezetimibe 10 mg vs Ezetimibe 10 mg in Subjects With Primary Dyslipidemia
Brief Title: Efficacy of Lapaquistat Acetate Alone and With Ezetimibe in Subjects With Primary Dyslipidemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475/EC303; 2005-002315-25 (EudraCT Number); U1111-1122-8322 (Registry Identifier: WHO)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lapaquistat Acetate 100 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Lapaquistat Acetate 100 mg QD + Ezetimibe (Experimental)
  Interventions: Drug: Lapaquistat acetate and ezetimibe
- Ezetimibe (Active Comparator)
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Lapaquistat acetate — Lapaquistat acetate 100 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD
Drug: Lapaquistat acetate and ezetimibe — Lapaquistat acetate 100 mg, tablets, orally, once daily and stable ezetimibe therapy for up to 24 weeks.
  Other Names: TAK-475; Zetia
  Arms: Lapaquistat Acetate 100 mg QD + Ezetimibe
Drug: Ezetimibe — Lapaquistat acetate placebo-matching tablets, orally, once daily and stable ezetimibe therapy for up to 24 weeks.
  Other Names: Zetia
  Arms: Ezetimibe

SUMMARY:
The purpose of the study is to determine the efficacy of lapaquistat acetate, once daily (QD), taken with ezetimibe on cholesterol levels in subjects with primary dyslipidemia

DETAILED DESCRIPTION:
In humans, cholesterol is acquired from dietary sources and is produced de novo in the liver, intestine, and various other tissues. Normally, the balance among cholesterol synthesis, dietary intake, and degradation is adequate to maintain healthy cholesterol plasma levels; however, in subjects with hypercholesterolemia, elevation in low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls (atherosclerosis) and subsequent coronary heart disease. Thus, it has been established that lowering the low-density lipoprotein cholesterol plasma concentrations effectively reduces cardiovascular morbidity and mortality. Additional lipid risk factors for coronary heart disease include elevated triglyceride, very low-density lipoprotein cholesterol and low-density lipoprotein cholesterol levels, and low levels of high-density lipoprotein cholesterol.

Despite changes in lifestyle and the availability of potent lipid-lowering agents, cardiovascular disease continues to be the major cause of death in Western Europe and North America. Serum cholesterol levels exceeding 5 mmol/L (193 mg/dL) are common in adults in Britain and much of Europe, the United States, Australia, and New Zealand, representing a serious public health concern.

Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (ie, statins) are the first-line monotherapies prescribed for the treatment of dyslipidemia, after diet and therapeutic lifestyle changes alone fail to reduce low-density lipoprotein cholesterol to desired levels. Statins reduce low-density lipoprotein cholesterol and triglycerides, increase high-density lipoprotein cholesterol, and improve endothelial function. Treatment with statins reduces the risk of a vascular event by about 30% in subjects with and without symptoms of arteriosclerosis; however, many subjects fail to reach recommended levels of low-density lipoprotein cholesterol reduction after receiving low-dose statins as a monotherapy. Consequently, the dosage of statins is often increased or an additional treatment is added; the latter has become an important therapeutic option for achieving increasingly stringent lipid targets set forth by international therapeutic guidelines.

Ezetimibe is a lipid-lowering compound that selectively inhibits intestinal absorption of cholesterol at the brush border of the small intestine, leading to a decrease in the delivery of intestinal cholesterol to the liver. Ezetimibe does not affect the absorption of triglycerides, fatty acids, bile acids, progesterone, ethinylestradiol, or fat-soluble vitamins A and D.

TAK-475 (lapaquistat acetate) is a squalene synthase inhibitor currently under development at Takeda for the treatment of dyslipidemia. This study will evaluate the efficacy and safety of lapaquistat acetate taken with ezetimibe in subjects with hypercholesterolemia. Total participation time in this study is expected to be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception from screening throughout the duration of the study and for 30 days following the last dose.
* Has a documented history of dyslipidemia with or without cardiovascular risk factors but without type 1 or 2 diabetes.
* At Randomization, participants must fulfill the above criteria and also have a mean fasting low density lipoprotein cholesterol levels greater than or equal to 3.36 mmol/L and less than or equal to 5.6 mmol/L and mean triglyceride levels less than or equal to 4.52 mmol/L.
* Is willing and able to comply with the recommended, standardized diet.

Exclusion Criteria:

* Has active liver disease or jaundice.
* Has a history of cancer, other than basal cell carcinoma, that had been in remission for less than 5 years prior to the first dose of study drug.
* Has an endocrine disorder, such as Cushing Syndrome, hyperthyroidism, or inappropriately treated hypothyroidism affecting lipid metabolism.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody, as determined by medical history and/or the subject's verbal report.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications, as determined by medical history and/or the subject's verbal report. .
* Has participated in any other clinical studies with lapaquistat acetate, was concurrently participating in another investigational study, had participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* Has a known hypersensitivity or history of intolerance to lapaquistat acetate or ezetimibe.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known Type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain and/or discontinuation of HMG-CoA reductase inhibitors due to myalgia at any time.
* Has uncontrolled hypertension despite medical treatment.
* Has inflammatory bowel or any other malabsorption syndrome or had had gastric bypass surgery or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of high alcohol intake within the previous 2 years.
* Has any other serious disease or condition at Visit 1 or Randomization that might reduce life expectancy, impaired successful management according to the protocol, or make the participant unsuitable to receive study drug.
* Has a history of coronary heart disease or coronary heart disease-risk factors comprised of:

  * Diabetes mellitus type 1 or 2
  * History or presence of myocardial infarction, angina pectoris, unstable angina, coronary angioplasty, coronary or peripheral arterial surgery (bypass graft), aortic aneurysm, transient ischemic attacks, or cerebrovascular accident;
  * Multiple risk factors that confer a 10-year risk of coronary heart disease greater than 20% based on the Framingham risk score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1267 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma Low Density Lipoprotein cholesterol | Week 24 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Triglycerides | Week 24 or Final Visit
Change from Baseline in Total Cholesterol | Week 24 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 24 or Final Visit
Change from Baseline in apolipoprotein B | Week 24 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 24 or Final Visit
Best corrected visual acuity | Week 24 or Final Visit
Adverse Events | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Clinical Laboratory Tests | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Vital Signs | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
12-lead Electrocardiogram | Weeks 12 and 24 or Final Visit
Physical Examination | Week 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (9):
- Estonia (2):
  - Tallinn
  - Tartu
- Riga, Latvia
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tyumen
- Kragujevac, Serbia

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985